CLINICAL TRIAL: NCT04635488
Title: Radiomics-based Prediction Model for Lateral Lymph Node Metastasis in Rectal Cancer
Brief Title: Prediction Model for Lateral Lymph Node Metastasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ziqiang Wang,MD, MD, West China Hospital
Other Study IDs: LLNM-2020
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; lymph node metastasis; prediction model
MeSH Terms: conditions — Rectal Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trainning group: 70% of the whole participants would be randomly divided into the training group to build the predicition model.
  Interventions: Procedure: lateral lymph node dissection
- validation group: 30% of the whole participant would be divided into the validation group to validate the model
  Interventions: Procedure: lateral lymph node dissection

INTERVENTIONS:
Procedure: lateral lymph node dissection — All participted would receive lateral lymph node dissection for rectal cancer.

SUMMARY:
Mid to low-lying rectal cancer patient with enlarged lateral lymph node befor treatment and receiving lateral lymph node dissection would be enrolled. Radiomics parameters of lateral lymph nodes would be extracted by expert software. Then a part of the nodes would be used as the training set to build the prediction model, and the another part nodes would be used as the validation set.

DETAILED DESCRIPTION:
After performing lateral lymph node dissection for the enrolled patients, we would find the targeted lateral node which was matched with the enlarged one in imaging from the specimen. Then the nodes would be send for pathological examination. Then we would extract the radiomics parameters of the nodes from the pretreatment CT and MRI with ITK-SNAP software. According to the pathological status, lymph nodes and corresponding radiomics parameters would be divided into positive and negative groups. Then significant parameters would be selected by R software. Then the prediction model with nomogram would be developed. 70% nodes would be used for for model development and the other 30% would be used for validation.

ELIGIBILITY:
Inclusion Criteria:

* middle to low-lying rectal adenocarcinoma patients with enlarged lateral lymph node ≥5mm for short diameter in CT and/or MRI

Exclusion Criteria:

* other kind of rectal tumor including neuroendocrine and malignant.
* high location rectal cancer.
* recurrent rectal cancer

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with rectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
metastasis rate of lateral lymph node | 2020.1-2022.12.31

CONTACTS AND LOCATIONS:
Locations (1):
- Guoxue Road 37#,West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
individual participant data (IPD) would not be available to other researchers.